CLINICAL TRIAL: NCT00214227
Title: ATM Variants in Radiotherapy
Brief Title: ATM Variants in Radiotherapy Patients
Status: Completed | Type: Observational
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Other Study IDs: RO05305; 2005-0122 (Other: Institutional Review Board); A533300 (Other: UW Madison); SMPH/HUMAN ONCOLOGY (Other: UW Madison)
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Last update posted 2019-11-19 (Actual); Status verified 2013-06

CONDITIONS: Radiotherapy
Keywords: patient who will undergo definitive radiotherapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — direct sequence analysis of all exons and intron-exon junctions of the ATM gene. DNA will be isolated from lympocytes using the PAX blood DNA system.

SUMMARY:
The purpose of this study is to compare the baseline incidence of variant alleles in the ATM and/or other DNA repair genes present in the Native American population versus the non-Native American population. It is thought that a higher baseline incidence of the variant alleles in the ATM gene may correlate to higher rates and higher grades of radiation toxicities noted in the Native American population.

ELIGIBILITY:
Inclusion Criteria:

* Indication for radiotherapy.
* Ability or desire to donate a blood sample and be followed closely for radiation toxicities

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who have been enrolled on RO02803.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2007-12; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
to determine baseline incidence of variant alleles in ATM | one blood draw
  to determine the baseline incidence of variant alleles in ATM resent in the population of Native americans with cancer who are undergoing radiation therapy to a similar group of non-native americans who have undergone or are undergoing raditohterapy

SECONDARY OUTCOMES:
to compare the baseline incidence of variant alleles in ATM | one blood draw
  to compare the baseline incidence of variant alleles in ATM resent in the population of Native americans with cancer who are undergoing radiation therapy to a similar group of non-native americans who have undergone or are undergoing raditohterapy

CONTACTS AND LOCATIONS:
Overall Officials: Mark Ritter, MD, PhD, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin Hospital and Clinics, Madison, Wisconsin, United States

REFERENCES:
- See also: University of Wisconsin Carbone Cancer Center — https://cancer.wisc.edu